CLINICAL TRIAL: NCT03962959
Title: Enhancement of Hippocampal Plasticity Using Repetitive Transcranial Magnetic Stimulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Arizona (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1812171968; R01AG062543 (NIH)
Record Dates: First submitted 2019-01-14; First posted 2019-05-24 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Mild Cognitive Impairment
Keywords: Mild Cognitive Impairment; Transcranial Magnetic Stimulation
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Excitatory TBS (Experimental): Excitatory TBS
  Interventions: Device: TBS
- Inhibitory TBS (Experimental): Inhibitory TBS
  Interventions: Device: TBS
- Sham TBS (Placebo Comparator): Sham TBS
  Interventions: Device: TBS

INTERVENTIONS:
Device: TBS — TMS is a non-invasive brain stimulation technique. The primary aim of the study will be to verify the deliverability of the TMS effect on the hippocampus and determine which stimulation protocol is more beneficial to each participant.
  Other Names: Theta Burst Stimulation (TBS)

SUMMARY:
The ultimate goal of this study is to develop non-invasive, painless repetitive transcranial magnetic stimulation (rTMS) protocols to prevent cognitive decline in patients with mild cognitive impairment (MCI) and cognitively normal individuals at high risk of developing Alzheimer's disease (AD). Currently, 1 in 9 adults over the age of 65 have AD, which currently totals more than 5 million Americans and this number is expected to rise as high as 16 million by 2050.

MCI is a clinical syndrome that represents the gray area between healthy aging and dementia. Those with amnestic MCI (aMCI) have memory problems more severe than normal for their age and education, but their symptoms are not as severe as those of people with AD. Patients with aMCI are at high risk for AD. Notably, roughly half of those with MCI will continue to progress and convert to clinical dementia within 3 years. Alternatively, it is also worthwhile to study cognitively healthy older adults who carry genes that may increase the risk of AD. The frequency of the human APOE gene ε4 allele increases in patients with AD and the ε4 allele is also associated with an earlier age of disease onset.

Currently, there are no known therapies that can effectively modify the progression and hallmark symptoms of AD. Therefore, it is crucial to provide an early intervention in patients with aMCI to delay or prevent the progression to AD.

More specifically, this project has two specific aims:

1. To plan personalized non-invasive brain stimulation location by brain Imaging with Magnetic Resonance Imaging (MRI) in Mild Cognitive Impairment (MCI)
2. To identify potential personalized cognitive enhancement strategy (such as dosage or patterns) of Transcranial Magnetic Stimulation (TMS) in MCI.

Techniques to artificially and precisely stimulate brain tissue are increasingly recognized as valuable tools both in clinical practice and in cognitive neuroscience studies among healthy individuals and people with clinical conditions. With these practices, researchers can safely stimulate specific regions of the brain to explore causal relationships that comprise the brain's circuitry and modulate behavior.

DETAILED DESCRIPTION:
In total, 60 participants (50-80 years old) with MCI will be recruited to participate in this trial.

Participants will be asked to receive 30 intervention sessions for three different protocols (10 sessions for each). Before and after the interventions, MRI and Cognitive tasks will be utilized again as the outcome measurements. There is a one-month interval between each protocol. Each intervention will be around half hour to an hour and each outcome measurement will take another two hours.

Each block includes:

* MRI+ Memory pre-assessment (2 hours/session)
* TMS * 10 (10 sessions; 0.5 hours/session)
* MRI+ Memory post-assessment (2 hours/session) Participants will experience each of the three TMS protocols. The total time commitment across these sessions will be approximately 27 hours.

There will be another 2 testing sessions to evaluate intervention effects. They will be scheduled at the beginning, and 1 month after the end of the intervention sessions. All sessions will take place in the Biosciences Research Laboratories (BSLR) Building (1230 N. Cherry Ave., Tucson, AZ 85721). The schematic below outlines the components of the sessions.

The investigators will acquire the following data during components for primary outcome measures and secondary measures.

1) Brain imaging data 2) Neuropsychological data and demographic data 3) Cognitive tasks 4) Biological sample

ELIGIBILITY:
Individuals with mild cognitive impairment (MCI Group)

Inclusion Criteria:

* Age 50-80 years
* MCI clinical criteria: (a) self- or informant-reported cognitive complaint; (b) preserved independence in functional abilities; and (c) absence of dementia.
* Objective cognitive impairment supported by the following measures of general cognitive function: (a) Mini-Mental State Exam (MMSE) 24-27 (inclusive); (b) Montreal Cognitive Assessment (MoCA) 18-26 (inclusive); or (c) Clinical Dementia Rating Scale score of 0.5.
* Right handed
* English speaking
* Able to attend daily intervention (Monday-Friday) for 4 weeks
* Not enrolled in another interventional study within 6 months prior to beginning this study

Exclusion Criteria:

* Contraindications to transcranial magnetic stimulation (TMS) or magnetic resonance imaging (MRI)
* Other neurological disorders (e.g. stroke, head injuries, or multiple sclerosis)
* Untreated depression
* Current cancer treatment or other medical problems that might independently affect cognitive function
* Clinical Dementia Rating Scale score more than 1.0

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-10-21 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Brain imaging data | Baseline
  The investigators will acquire MRI images to measure structural and functional connectivity, respectively.
NACC Neuropsychological batteries | Baseline
  The investigators will use Neuropsychological batteries, which would calculate the Z-score, for measuring cognitions. With Z-score, the investigators can classify participants into MCI or non-MCI group.
Correction rate in memory association recall | Baseline
  Memory tasks will be implemented and measure the correct rate to assess memory function.
Specimen sample | 1 day (Only once in the beginning phase)
  A specimen for DNA will be collected and determine whether participants have APOE genotype.

SECONDARY OUTCOMES:
Brain imaging data | 2 weeks after the intervention phase begin
  The investigators will acquire MRI images to measure structural and functional connectivity, respectively.
Correction rate in memory association recall | 2 weeks after the intervention phase begin
  Memory tasks will be implemented and measure the correct rate to assess memory function.

OTHER OUTCOMES:
Brain imaging data | an average of 1 month
  The investigators will acquire MRI images to measure structural and functional connectivity, respectively.
Brain imaging data | 3 months after the intervention phase complete
  The investigators will acquire MRI images to measure structural and functional connectivity, respectively.
NACC Neuropsychological batteries | an average of 1 month
  The investigators will use Neuropsychological batteries, which would calculate the Z-score, for measuring cognitions function. With Z-score, the investigators can classify participants into MCI or non-MCI group.
NACC Neuropsychological batteries | 3 months after the intervention phase complete
  The investigators will use Neuropsychological batteries, which would calculate the Z-score, for measuring cognitions. With Z-score, the investigators can classify participants into MCI or non-MCI group.
Correction rate in memory association recall | an average of 1 month
  Memory tasks will be implemented and measure the correct rate to assess memory function.
Correction rate in memory association recall | 3 months after the intervention phase complete
  Memory tasks will be implemented and measure the correct rate to assess memory function.

CONTACTS AND LOCATIONS:
Locations (1):
- Bioscience Research Laboratory, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No